CLINICAL TRIAL: NCT01170741
Title: A Tailored Cue Card HIV/STI Intervention for High Risk Groups Pilot Study
Brief Title: Computer-Assisted Tailored Cue-card Health [CATCH] Study
Acronym: CATCH
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: RTI International (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1R21DA026771 (NIH)
Record Dates: First submitted 2010-07-26; First posted 2010-07-27 (Estimated); Last update posted 2012-10-25 (Estimated); Status verified 2012-10

CONDITIONS: Human Immunodeficiency Virus; STDs; Hepatitis, Viral, Human
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Sexually Transmitted Diseases; Hepatitis, Viral, Human

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Delayed Control Condition (No Intervention): Participants assigned to the delayed treatment control condition will be offered biological testing and the tailored cue-card intervention upon completion of their 3- month follow-up interview. Use of a delayed treatment control group design will permit us to separate intervention effects on HIV risk behaviors from the general effects of participating in the study and completing a detailed HIV risk assessment.
  Interventions: Behavioral: Tailored Cue Cards

INTERVENTIONS:
Behavioral: Tailored Cue Cards — The proposed intervention uses education to increase knowledge and skill building to influence behavior-specific self-efficacy and outcome expectations. In addition to providing general information regarding drug use and diseases, the cue-cards include information that is designed to raise awareness regarding perceived threats (perceived susceptibility and perceived severity) related to HIV and other STIs and blood-borne infections, which increases motivation to reduce risk behaviors. The cue-cards also provide information regarding risk reduction strategies. The cue-cards also contain instructions on how to anticipate and avoid risky situations (e.g., using alcohol or drugs prior to sex). This information is augmented with an exercise that involves modeling and guided practice. This combination of information and exercises modifies outcome expectations by increasing confidence (i.e., perceived self-efficacy) that a protective action can be performed

SUMMARY:
This study will draw from proven interventions to refine and pilot test a cue card driven computer-assisted intervention, along with HIV/STI testing, that will be tailored to each participant's demographic characteristics, risk behaviors, and biological test results. The specific aims of the proposed study are:

1. To refine a cue card driven computer-assisted risk reduction intervention that will be tailored to each participant's demographic characteristics (e.g., gender, ethnicity), risk behaviors, and biological test results (HIV, hepatitis B and C, syphilis and herpes).
2. To pilot test the tailored intervention's effects on sexual risk behaviors (e.g., frequency of unprotected sex, condom use), drug use during sex and injection risk behaviors (e.g., direct syringe sharing, indirect sharing practices) using a two-group randomized design that compares the tailored intervention with a delayed treatment control condition.
3. To assess the feasibility and acceptability of the tailored intervention in a rural setting.

ELIGIBILITY:
Inclusion Criteria:

The sample of 120 will be drawn from the Raleigh-Durham, NC metro area with the following targets:

* 40 MSM (at least 12 African American, 12 non-Hispanic white and 12 Hispanic) - eligibility includes unprotected sex with another male in the past 30 days
* 40 sex workers (at least 6 male and 6 female of each race/ethnicity) - eligibility includes unprotected sex within the last 30 days and exchange of sex for money or drugs within the past 30 days
* 40 drug users who are not sex workers or MSM (at least 2 males and 2 females of each race/ethnicity) - eligibility includes use of methamphetamine, crack or powder cocaine, or heroin in the past 30 days and unprotected intercourse and/or syringe sharing in the past 30 days.

Additional eligibility criteria include the following:

* be 18 years of age or older
* self-identify as male or female
* self-identify as African American, non-Hispanic white or Hispanic
* not currently be in or seeking substance use treatment
* speak and understand written English proficiently
* be a resident of Wake, Durham, Orange, Johnston or Chatham counties, with no plans to move in the next 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2010-06; Primary Completion 2011-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Sex risk | 3 months
  Compared with participants assigned to the control condition, participants assigned to the tailored intervention will report lower rates of unprotected sex at 3-month follow-up.

SECONDARY OUTCOMES:
Injection risk | 3 months
  Compared with IDU participants assigned to the control condition, IDU participants assigned to the tailored intervention will report lower rates of direct and indirect syringe sharing at 3-month follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: William A Zule, DrPH, Principal Investigator — RTI International
Locations (1):
- RTI International - Wake County Field Site, Raleigh, North Carolina, United States